CLINICAL TRIAL: NCT01405846
Title: Tyrosine Kinase Inhibitors in DyplAsia of Lung Epithelium
Brief Title: Feasibility Study to Estimate Number of Patients With Precancerous Areas in Their Airways and the Response to Gefitinib
Acronym: TIDAL1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: AstraZeneca (Industry); Noble Organisation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01425; 2010-023355-29 (EudraCT Number); 11/H0304/8 (Other: Research Ethics Committee)
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer; Head and Neck Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib (Other): Single arm study
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250mg od for 6 months
  Other Names: IRESSA

SUMMARY:
We are going to use a special type of bronchoscopy test to examine patients who have had previous surgical treatment for lung cancer or head and neck cancer. The aim is to determine a) whether we can identify precancerous changes in their airways b) whether this type of testing is acceptable and c) get an initial idea of whether a new drug called gefitinib has any effect on precancerous areas in the airway.

ELIGIBILITY:
* Age 18 years or above
* Resected NSCLC or Squamous cell Head & Neck cancer treated curatively
* All treatment, including any adjuvant treatment with radiotherapy and/or chemotherapy completed at least 3 months prior to study entry
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
* Suitable for flexible bronchoscopy
* Able to give signed informed consent
* Adequate haematological, kidney and liver function:

  * Serum alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN)
  * Total serum bilirubin ≤1.5 x ULN
  * Absolute neutrophil count (ANC) ≥1500/μL
  * Platelets ≥100,000/μL
  * Haemoglobin ≥9.0 g/dL
  * Sufficient renal function to allow administration of contrast medium (in line with Royal College of Radiologists guidelines).

In addition, the following inclusion criteria must be met during the screening period in order to confirm eligibility for the study treatment

* No evidence of malignant disease activity on screening
* High grade dysplasia on autofluorescence bronchoscopy analysis
* No evidence of pulmonary fibrosis or interstitial lung disease on screening CT

Exclusion Criteria:

* Diagnosis of any second malignancy within the 5 years from date of enrolment, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix uteri that has been adequately treated with no evidence of recurrent disease for 12 months
* Evidence of severe or uncontrolled systemic disease or psychiatric disorder that would interfere with the patient's safety
* Known severe hypersensitivity to Gefitinib or any of the excipients of the product
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease
* Pre-existing idiopathic pulmonary fibrosis
* History of allergy to contrast medium
* Insufficient lung function as determined by either clinical examination or an arterial oxygen tension (PaO2) of < 9.3kpa
* Inability to swallow oral medications
* Presence of active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhoea or any condition which would interfere with absorption of an oral drug.
* Past medical history of keratitis
* Past medical history of Sjogren's syndrome
* Pregnant or breast-feeding
* Male and female patients (of childbearing age) not using, or not willing to use, protocol mandated contraception
* Prior EGFR inhibitor use.
* Concurrent medication with known potent CYP3A4 inhibitors and inducers and/or dosing within 7 days of date of enrolment (e.g.. ketoconazole, rifampin, phenytoin, carbamazepine, barbiturates or herbal preparations containing St John's wort/Hypericum perforatum etc.) or use of other concomitant medication incompatible with study drug (see SmPC)
* Current treatment on another therapeutic clinical trial or previous investigational agent in the last 12 weeks (supportive care trials or non-treatment trials are allowed)
* Previous enrolment or treatment in the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of high grade dysplasia of the bronchial epithelium in patients at high risk of lung dysplasia | during the screening broncoscopy - carried out within the first month post consent
  Patients will have white/blue light bronchoscopy with biopsy of identified lesions. The incidence of high grade lung epithelial dysplasia will be recorded.

SECONDARY OUTCOMES:
Acceptability of screening patients as measured by success of trial recruitment | 12 months
Response of high grade dysplasia to treatment (complete / partial / stable / progression) | 6 & 12 months
  To be estimated by photography & biopsy of the lesions & comparison with previous findings:
  Complete response: Complete resolution of a dysplastic lesion Partial response: Reduction of a dysplastic lesion by >=50% OR Reduction in grade of a high grade dysplastic lesion Progressive disease: Development of a new area of high grade dysplasia or invasive malignancy in an area of previous low grade dysplasia or normal epithelium OR Development of a higher grade lesion in an area of previous high grade dysplasia OR Increase in surface area of >=50%.
  Stable disease: None of the above.
Toxicity and acceptability of treatment (proportion of patients refusing study entry). | 2 weeks, 4 weeks, 3 & 6 months
Successful biobanking of samples | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim Eisen, Professor, Study Chair — Papworth Hospital NHS Trust; Robert Rintoul, Dr, Principal Investigator — Papworth Hospital NHS Trust
Locations (1):
- Papworth Hospital NHS Trust, Papworth Everard, Cambs, United Kingdom